CLINICAL TRIAL: NCT06263738
Title: Cold and Heat Investigation to Lower Levels of Depression
Acronym: CHILL'D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barry Sandler (Other)
Collaborators: Steadman Philippon Research Institute (Other)
Responsible Party: Sponsor-Investigator, Barry Sandler, Medical Director of Vail Healthspan, Vail Health Behavioral Health
Organization: Vail Health Behavioral Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20244106
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Depression; Mood Disorders; Healthy (Controls)
Keywords: Depression; Mood Disorders; Mental Health; Integrative Health; Hyperthermia; Sauna; Cold Plunge
MeSH Terms: conditions — Depression; Mood Disorders; Psychological Well-Being; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants who meet inclusion/exclusion criteria will be stratified by use of antidepressant medication and randomized with a 1-to-1 allocation to receive a single session of WBH or a single session of WBH followed immediately by cold plunge (WBH+cold).
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary outcome data will be collected by trained raters blinded to participant group assignment and study visit number. The participant will be blinded to their treatment assignment until the end of the WBH treatment, at which point they will be directed to either complete a cool-down period in the sauna device or proceed to the cold plunge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Depression + Whole Body Hyperthermia (Active Comparator): Participants experiencing depression will receive a single heat treatment using the Clearlight Sauna Dome lasting up to 140 minutes.
  Interventions: Procedure: Whole Body Hyperthermia
- Depression + Whole Body Hyperthermia + Cold Water Plunge (Active Comparator): Participants experiencing depression will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes followed by a cold plunge session lasting up to 10 minutes.
  Interventions: Procedure: Whole Body Hyperthermia; Procedure: Cold Water Plunge
- No Depression + Whole Body Hyperthermia (Active Comparator): Participants not experiencing depression will receive a single heat treatment using the Clearlight Sauna Dome lasting up to 140 minutes.
  Interventions: Procedure: Whole Body Hyperthermia
- No Depression + Whole Body Hyperthermia + Cold Water Plunge (Active Comparator): Participants not experiencing depression will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes followed by a cold plunge session lasting up to 10 minutes.
  Interventions: Procedure: Whole Body Hyperthermia; Procedure: Cold Water Plunge

INTERVENTIONS:
Procedure: Whole Body Hyperthermia — Participants in the heat exposure alone group will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes
  Other Names: Infrared Sauna; Whole Body Heating
Procedure: Cold Water Plunge — Participants in the heat exposure and cold plunge group will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes followed by a cold plunge session in 55 degree (Fahrenheit) water, lasting up to 10 minutes.
  Other Names: Cold Plunge; Cold Water Exposure
  Arms: Depression + Whole Body Hyperthermia + Cold Water Plunge; No Depression + Whole Body Hyperthermia + Cold Water Plunge

SUMMARY:
This study will recruit 112 medically healthy adults (aged 18-65) currently experiencing depressive symptoms to be randomized to receive either a single Whole Body Hyperthermia (heat therapy) treatment or a Whole Body Hyperthermia treatment followed by a cold water plunge. Participants will complete a baseline assessment of their depressive symptoms as well as 1-week and 2-week post-treatment followup assessments.

DETAILED DESCRIPTION:
The CHILL'D Study aims to figure out how using heat exposure as a treatment for major depressive disorder (MDD) can work better. The researchers want to see if being exposed to heat followed by cold plunge can help people feel better emotionally compared to just being exposed to heat alone.

To answer study questions, 112 adults, ages 18 to 65 experiencing depression for at least 60 days and who meet study eligibility criteria, will be randomized with 1-to-1 allocation to receive either 1) a single session of heat exposure or 2) a single session of heat exposure followed immediately by cold plunge.

A second cohort of up to 50 adults, ages 18 to 65 not experiencing MDD will be randomized with 1-to-1 allocation to the same interventions.

Participants in the heat exposure alone group will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes. Participants in the heat exposure and cold plunge group will receive a single heat session using the Clearlight Sauna Dome lasting up to 140 minutes followed by a cold plunge session lasting up to 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who currently meet study criteria for depression or individuals who do not currently meet criteria for depression
* English or Spanish speaking (able to provide informed consent and complete questionnaires in one of these languages)
* Able and willing to adhere to trial requirements, including attending all trial visits, preparatory and follow-up sessions, and completing all trial evaluations.

Exclusion Criteria:

* Previous adverse reaction to hypothermia, hyperthermia and/or infrared exposure
* Use of any medication that may impact thermoregulatory capacity.
* Pregnancy, active lactation, or intention to become pregnant during the study period.
* Endorses current active suicidal ideation with a plan or made a suicide attempt in the prior 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline/Treatment (Visit 1), 1 Week Post-Treatment (Visit 2), 2 Weeks Post-Treatment (Visit 3)
  The MADRS is a validated 10-item questionnaire to assess depression severity and is commonly used to assess efficacy of an intervention in clinical trials. Each item of the MADRS is measured on a scale of 0 to 6 (for a total score of 0 to 60) with higher scores indicating more severe depression. The MADRS includes questions on the following symptoms: 1. Reported sadness; 2. Apparent sadness; 3. Inner tension; 4. Reduced sleep; 5. Reduced appetite; 6. Concentration difficulties; 7. Lassitude; 8. Inability to feel; 9. Pessimistic thoughts; 10. Suicidal thoughts. Items are scored via a clinical interview that progresses from more broadly phrased questions about symptoms to more detailed queries that allow a precise rating of severity.

SECONDARY OUTCOMES:
Warwick Edinburgh Mental Well-Being Scale (WEMWBS) | Baseline/Treatment (Visit 1), 1 Week Post-Treatment (Visit 2), 2 Weeks Post-Treatment (Visit 3)
  The WEMWBS was designed to measure the psychological well-being of a population and has been shown to be responsive to novel interventions such as psychedelics. WEMWBS has 14 questions scored using a five-point Likert scale. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing. Items on the questionnaire are rated on a 5-point scale, where 1= "None of the time", 2= "rarely", 3= "some of the time", 4= "often", 5= "all the time". Scores reflect feelings and thoughts in the two weeks prior to answering the questionnaire. The WEMWBS assesses both emotional and functional aspects of mental well-being. Total scores range from 14 to 70, with higher scores correlating to higher levels of well-being.
Patient Reported Outcome Measure Information System (PROMIS) 8A - Anxiety | Baseline/Treatment (Visit 1), 1 Week Post-Treatment (Visit 2), 2 Weeks Post-Treatment (Visit 3)
  The PROMIS Anxiety measure focuses on fear (e.g., worry, feelings of panic), anxious misery (e.g., dread), hyperarousal (e.g., tension, nervousness, restlessness), and somatic symptoms related to arousal (e.g., cardiovascular symptoms, dizziness) and has been found to be a clinically validated measure of anxiety. The PROMIS 8A--Anxiety is comprised of eight items, each rated on a scale from 1 ("Never") to 5 ("Always"). Total scores range from 8 to 40, with higher scores correlating to higher levels of anxiety.
Sheehan Disability Scale (SDS) | Baseline/Treatment (Visit 1), 1 Week Post-Treatment (Visit 2), 2 Weeks Post-Treatment (Visit 3)
  The SDS is a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in the patient's life are impaired by psychiatric symptoms, including depression. This scale has been used widely in psychopharmacology randomized, controlled trials and has been accepted by the Food and Drug Administration (FDA) for functional disability labeling. The SDS uses visual-spatial, numeric, and verbal descriptive anchors simultaneously to assess disability across 3 domains: work, social life, and family life. The SDS asks participants to rate the extent to which their 1) work/school, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analogue scale. Total scores range from 0 to 30, with higher scores correlating to higher levels of disability.
Quality of Life Enjoyment & Satisfaction Questionnaire Short Form (Q-LES-Q SF) | Baseline/Treatment (Visit 1), 1 Week Post-Treatment (Visit 2), 2 Weeks Post-Treatment (Visit 3)
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form version contains 16 items assessing changes in quality of life, divided into the following sections: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. A total score is derived from summing the first 14 items on the scale, with the last 2 items serving as stand-alone queries. Total score ranges from 14 to 70, with higher scores correlating with higher levels of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Sandler, DO, Principal Investigator — Vail Health Behavioral Health
Locations (1):
- Vail Health Behavioral Health Innovation Center, Edwards, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including, but not limited to, demographics, questionnaires, and adverse events will be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Following publication of primary study findings.
Access Criteria: De-identified data will be made available to qualified researchers in a way that protects subject confidentiality and adheres to HIPAA policies. Both internal and external requests for data will be handled by the study team to ensure equitable access, fairness, and safeguards. After reviewing a short proposal prepared by an external investigator, the study team will approve requests with appropriate experimental design, scientific merit, and Institutional Review Board (IRB) approval and recommend revisions for proposals requiring further justification or modifications. Informed consent documents will provide sufficient detail about the intent to archive, share, and re-analyze data.